CLINICAL TRIAL: NCT05075837
Title: Virus-specific T-cell Immunity for the Treatment of Some Resistant Viral Infections After Allogeneic Hematopoietic Stem Cell Transplantation(HSCT)
Brief Title: Adoptive T-cell Therapy for Resistant Viral Infections After Allogeneic HSCT
Acronym: VS-TC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Maura Faraci, Principal investigator, Istituto Giannina Gaslini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGianninaGaslini
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Viral Infection After HSCT
Keywords: CMV; adenovirus; EBV; adoptive T cell therapy; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Intervention Model Description: Phase I, open-label, single-arm, non-randomized study, monocentric.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virus-specific T cells for the treatment of active viral infections following allogeneic HSCT. (Experimental): Virus specific T lymphocytes selected in vitro from a family donor to treat some refractory viral infections as Adenovirus (ADV), Ebstein Barr virus (EBV), Cytomegalovirus (CMV) that developed in young patients (age between 0 and 21 years) after allogeneic hematopoietic cell transplantation (allo-HSCT)
  Interventions: Biological: Virus -specific T cells

INTERVENTIONS:
Biological: Virus -specific T cells — The product is obtained by leukapheresis of a family donor responsive to the virus: consists of virus- specific T lymphocytes (both CD4+ and CD8+) resuspended in PBS / EDTA buffer plus 0.5% Albumin Human. The productive process lasts two consecutive days and includes two phases: a brief activation with specific viral peptide followed by immunomagnetic separation using the CliniMACS® CCS (IFNγ) capture system which allows a fast and automated separation of IFNγ secreting lymphocytes

SUMMARY:
The aim of the study is to evaluate the adverse events and the efficacy of virus specific T lymphocytes selected in vitro from a family donor to treat some refractory viral infections as Adenovirus (ADV), Ebstein Barr virus (EBV), Cytomegalovirus (CMV) that developed in young patients (age between 0 and 21 years) after allogeneic hematopoietic cell transplantation (allo-HSCT) performed at the Transplant Clinical Unit of the IRCCS G. Gaslini Institute (IGG).

DETAILED DESCRIPTION:
The rationale for the study is based on the evidence that, despite the progress obtained in the management and prevention of viral infections in the patients who received allo-HSCT, some viral infections continue to be severe complications that may occurred before the immune recovery. Some of these viral reactivations are not responsive to the first or second line treatment and their treatment may be represent an important issue. The adoptive cellular immunotherapy based on the infusion of virus-specific T lymphocytes represent a valid therapeutic option and the quick access to this cellular therapy is crucial to prevent severe organ complications related to viral infection. In this study, the use of virus-specific T lymphocytes obtained from a seropositive family donor, briefly activated in vitro and immunomagnetically captured by their capacity to secrete IFN-gamma allows to obtain a rapidly usable T-lymphocyte population (both CD4+ and CD8+) potentially able to expand into the patient. The effectiveness, safety (peptides used are synthetic, no animal components, closed system production), good tolerance and speed of modality (less than 36 hours for production) is reported by many clinical studies.

ELIGIBILITY:
Inclusion criteria:

* Allogeneic transplant with any cells source and conditioning regimen
* Age between 0-21 years
* Viral infection/reactivation (CMV, EBV, ADV)
* Resistance of viral infections to treatments
* Absence of concomitant severe uncontrolled infections
* Life expectancy exceeding 30 days
* Absence of acute or chronic uncontrolled Graft versus Host Disease (GvHD)
* Absence of acute kidney damage (creatinine value> 3 times the value normal with respect to age) not related to viral infection;
* Absence of severe acute liver injury (direct bilirubin> 3mg / dl or glutamic-oxaloacetic transaminase -SGOT> 500 UI/L) not related to viral infection;
* Presence of informed consent to the treatment of the patient / parent /legal guardian.

Exclusion Criteria:

* Absence of a suitable donor (seronegativity for the virus in question and / or failure to respond to the secretion test)
* Patient with severe renal and/or hepatic impairment as specified above
* Primary or secondary graft failure
* Relapse of malignant underlying disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-27 (Estimated); Primary Completion 2024-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Adverse events | from day +1 of infusion until day +56
  To collect any adverse event defined as any significant alteration of vital signs and / or organ function, expressed in clinical, hematochemical and radiological findings according to version 5 of the Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Specific cell viral immunity | from day +1 of infusion until day +56
  To evaluate the specific cell viral immunity for some virus defined as presence and number of CD3 + IFN-gamma + lymphocytes count in the patient's peripheral blood
Variation of viremia | from day +1 of infusion until day +56
  To evaluate viremia variations with the measurement of viral PCR after the infusion of virus-specific T lymphocytes evaluated regularly 2 times a week.
Organ damage | from day +1 of infusion until day +56
  To report any clinical and/or laboratory changes related to the viral infection
Overall survival | from day +56 to 12 months
  To evaluate the overall survival (OS) after virus-specific T lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Maura Faraci, MD, Principal Investigator — Istituto G. Gaslini

IPD SHARING:
Plan to Share IPD: No
IPD are to be shared with hematologists and oncologists of our Institute